CLINICAL TRIAL: NCT06489548
Title: Assessment of Foralumab Safety and Modulation of Microglial Activation Evaluated by PET Imaging in Patients With Early Symptomatic Alzheimer's Disease
Brief Title: Assessment of Foralumab Safety and Modulation of Microglial Activation in Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Tiziana Life Sciences LTD (Industry)
Responsible Party: Principal Investigator, Gad A. Marshall, MD, Director of Clinical Trials, Center for Alzheimer Research and Treatment, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P003329; TILS-024 (Other: FDA)
Record Dates: First submitted 2024-05-28; First posted 2024-07-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dementia; Alzheimers Disease; Mild Cognitive Impairment Due to Alzheimer's Disease
Keywords: Alzheimers; Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: This cohort of subjects will receive 100µg/dosing day vs. placebo throughout the study. (Active Comparator): This group will receive a nasal spray three times a week for two weeks, followed by a one-week rest. That cycle will occur three more times for a total of three months of drug intervention.
  Interventions: Drug: Foralumab TZLS-401 100 µg
- Arm B: This cohort of subjects will receive 50µg/dosing day vs. placebo throughout the study. (Active Comparator): This group will receive a nasal spray three times a week for two weeks, followed by a one-week rest. That cycle will occur three more times for a total of three months of drug intervention.
  Interventions: Drug: Foralumab TZLS-401 50 µg

INTERVENTIONS:
Drug: Foralumab TZLS-401 50 µg — Foralumab is a nasal anti-CD3 antibody. It will be administered in doses of 50 µg vs. placebo.
  Arms: Arm B: This cohort of subjects will receive 50µg/dosing day vs. placebo throughout the study.
Drug: Foralumab TZLS-401 100 µg — Foralumab is a nasal anti-CD3 antibody. It will be administered in doses of 100 µg vs. placebo.
  Arms: Arm A: This cohort of subjects will receive 100µg/dosing day vs. placebo throughout the study.

SUMMARY:
This phase 2a study will research the safety and tolerability of Foralumab, a human anti-CD3 antibody. An antibody is a molecule secreted by the immune system. These molecules are created to identify a specific pathogen. Previous data on experimental mice has suggested that Foralumab increases the immune system activity in the brain to reduce the inflammation of microglia, the brain's main immune cells. This combination of increased immune reactivity and less microglia inflammation may improve the immune response throughout the brain. Alzheimer's disease and other forms of dementia are characteristically known for the build-up of certain proteins in the brain. This trial will evaluate whether nasal Foralumab can improve cognition in participants with mild cognitive impairment due to early Alzheimer's or dementia.

The trial will ask participants to administer Foralumab nasally three times a week for eight weeks. The administration will occur intermittently, with breaks between each dosing cycle. Participants will also receive brain scans (Amyloid PET and MRI), undergo cognitive testing, blood draws, and physical, neurological, and nasal exams. Volunteers are expected to remain in the trial for six months.

DETAILED DESCRIPTION:
Preliminary data has shown that Foralumab, a human anti-CD3 antibody, may improve cognition in APP/PS1and 3xTg mouse models of AD. Nasal Foralumab has been given to healthy volunteers with progressive multiple sclerosis (MS). When given nasally for five consecutive days, doeses up to 250 µg are well-tolerated.

This is a randomized, double-blind, placebo-controlled study assessing two dose levels of nasal foralumab (50 µg/dosing day and 100 µg/dosing day) or placebo, given in three-week "treatment cycles". A treatment cycle is defined as Investigational Product (IP) dosing on Monday, Wednesday, and Friday for two consecutive weeks, followed by a one-week pause in dosing or a "rest week." All treatment cycles follow the identical dosing regimen. Randomization will be 3:1 Active to Placebo.

Two cohorts of eight (8) subjects each will be enrolled in this study, and enrollment in these cohorts will be staggered. Both cohorts, Cohort A and Cohort B, will consist of six (6) subjects who will complete three months (4 cycles) of active treatment and two (2) subjects who receive Placebo treatment. Enrollment into Cohort B may begin once all subjects in Cohort A complete 2 cycles of treatment.

Subjects will be screened and enrolled at the Center for Alzheimer Research and Treatment (CART). Initial treatment visits will occur in the Center for Clinical Investigation (CCI) with follow-up visits occurring in CART. Both centers are in the Building for Transformative Medicine, Brigham and Women's Hospital (BWH) at 60 Fenwood Road, Boston, MA 02115.

Subjects will undergo screening procedures, including laboratory studies (hematology, clinical chemistry, CRP, EBV serology, HIV testing, Hepatitis B and Hepatitis C), vital signs, cognitive testing, and a complete physical exam by the physician investigator or a mid-level practitioner, and a detailed neurologic examination performed by a neurologist. Each subject must have normal laboratory tests, or results must be in a clinically acceptable range in the opinion of the Investigator. An additional screening visit will consist of an amyloid PET scan (if subjects do not already have those results prior to screening). Prior to each treatment cycle and at the end of treatment, an ENT physician will conduct a nasal exam and safety blood labs will be collected. At baseline and end of treatment, each subject will have blood samples collected for immunological study and undergo an MRI and a microglial PET scan. Blood samples for immunologic studies will be collected at baseline and after 3 months of treatment. A lumbar puncture will be performed at the screening visit and after 3 months of treatment to assess for changes in amyloid and tau.

ELIGIBILITY:
Inclusion Criteria:

1. The Sponsor will rely on NIA-AA Alzheimer's Disease Diagnostic Guidelines for Early Symptomatic Alzheimer's Disease (AD) with a 20-30 MMSE score, Clinical Dementia Rating (CDR) global score of 0.5 or 1, and impaired memory performance below an education adjusted cut-off score on the Logical Memory II subscale delayed paragraph recall (LM-IIa) of the Wechsler Memory Scale- Revised (WMS-R) (127) (≥16 years: ≤8; 8-15 years: ≤4; 0-7 years: ≤2).
2. Age between 60 and 85 years (inclusive).
3. Good general health with no disease likely to interfere with the study assessments.
4. On a stable medication regimen for eight weeks prior to the study and is anticipated to remain stable during the study.
5. Subject is not pregnant, lactating, or of childbearing potential (i.e., women must be two years post-menopausal or surgically sterile). If a woman is of childbearing potential, her partner must use barrier contraception throughout the study.
6. Amyloid-positive PET scan (performed only if the subject meets all other inclusion criteria). An amyloid-positive PET scan is classified by an SUVR composite score cutoff of 1.18 units. Prior evidence of amyloid positivity by PET or CSF will also be accepted for eligibility.
7. Ability to understand and provide informed consent.
8. Has availability of a study partner who has regular contact with the participant and knows him/her well.

Exclusion Criteria:

1. Any significant neurologic disease including Parkinson's disease, stroke, multiinfarct dementia, frontotemporal dementia, Lewy body dementia, normal pressure hydrocephalus, brain tumor, brain hemorrhage with persistent neurologic deficits, progressive supra-nuclear palsy, seizure disorder, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
2. Clinically significant or unstable medical conditions, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic diseases.
3. History of autoimmune disease.
4. Current treatment with immunomodulatory or immunosuppressive drugs or corticosteroid administration by any route of administration (including nasal corticosteroids) within the past month.
5. Major depressive disorder (within the past 1 year), or a history of bipolar disorder, or a history of schizophrenia.
6. History of alcohol or substance abuse or dependence within the past two years.
7. History of malignancy within the past 3 years.
8. Clinically significant abnormalities in screening laboratories (defined as greater than mild on the FDA's vaccine toxicity grading scale).
9. Participation in another clinical trial of an investigational drug concurrently or within the past 30 days.
10. Low affinity TSPO binders (for PET ligand [18F]PBR06) determined by having a Thr/Thr polymorphism in the TSPO gene at screening.
11. Sensitivity to florbetapir F18.
12. Active COVID-19 disease.
13. Amyloid-negative PET scan.
14. COVID-19 vaccine within the past ten days or any other vaccine within the past seven days (at dosing)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events in drug versus placebo groups. | From baseline to the end of study, up to 20 weeks.
  Establish the safety and tolerability of nasal foralumab dosing in subjects as a percentage of drug and placebo groups who experience adverse events.
Assessment of microglial function via PET scan using the ligand [18F]PBR06 | From baseline to end of study, up to 20 weeks.
  The ligand [18F]PBR06 provides a quantification of microglial activation during a PET scan. The investigatorshope to use this tracer at the start and end of the study to examine how the use of Foralumab may affect microglial function.
Measure the effect of foralumab on the ratio of CD4/CD8 memory/naïve T cells biomarkers in blood | From baseline to the end of treatment, up to 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alzheimer Research and Treatment, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou R, Ji B, Kong Y, Qin L, Ren W, Guan Y, Ni R. PET Imaging of Neuroinflammation in Alzheimer's Disease. Front Immunol. 2021 Sep 16;12:739130. doi: 10.3389/fimmu.2021.739130. eCollection 2021. PMID 34603323
- [Background] Wu HY, Quintana FJ, Weiner HL. Nasal anti-CD3 antibody ameliorates lupus by inducing an IL-10-secreting CD4+ CD25- LAP+ regulatory T cell and is associated with down-regulation of IL-17+ CD4+ ICOS+ CXCR5+ follicular helper T cells. J Immunol. 2008 Nov 1;181(9):6038-50. doi: 10.4049/jimmunol.181.9.6038. PMID 18941193
- [Background] Toly-Ndour C, Lui G, Nunes MM, Bruley-Rosset M, Aucouturier P, Dorothee G. MHC-independent genetic factors control the magnitude of CD4+ T cell responses to amyloid-beta peptide in mice through regulatory T cell-mediated inhibition. J Immunol. 2011 Nov 1;187(9):4492-500. doi: 10.4049/jimmunol.1003953. Epub 2011 Sep 26. PMID 21949026
- [Background] Sakaguchi S, Yamaguchi T, Nomura T, Ono M. Regulatory T cells and immune tolerance. Cell. 2008 May 30;133(5):775-87. doi: 10.1016/j.cell.2008.05.009. PMID 18510923
- [Background] Ogura M, Deng S, Preston-Hurlburt P, Ogura H, Shailubhai K, Kuhn C, Weiner HL, Herold KC. Oral treatment with foralumab, a fully human anti-CD3 monoclonal antibody, prevents skin xenograft rejection in humanized mice. Clin Immunol. 2017 Oct;183:240-246. doi: 10.1016/j.clim.2017.07.005. Epub 2017 Jul 21. PMID 28739191
- [Background] Moreira TG, Matos KTF, De Paula GS, Santana TMM, Da Mata RG, Pansera FC, Cortina AS, Spinola MG, Baecher-Allan CM, Keppeke GD, Jacob J, Palejwala V, Chen K, Izzy S, Healey BC, Rezende RM, Dedivitis RA, Shailubhai K, Weiner HL. Nasal Administration of Anti-CD3 Monoclonal Antibody (Foralumab) Reduces Lung Inflammation and Blood Inflammatory Biomarkers in Mild to Moderate COVID-19 Patients: A Pilot Study. Front Immunol. 2021 Aug 12;12:709861. doi: 10.3389/fimmu.2021.709861. eCollection 2021. PMID 34475873
- [Background] Mayo L, Cunha AP, Madi A, Beynon V, Yang Z, Alvarez JI, Prat A, Sobel RA, Kobzik L, Lassmann H, Quintana FJ, Weiner HL. IL-10-dependent Tr1 cells attenuate astrocyte activation and ameliorate chronic central nervous system inflammation. Brain. 2016 Jul;139(Pt 7):1939-57. doi: 10.1093/brain/aww113. Epub 2016 May 31. PMID 27246324
- [Background] Kuhn C, Weiner HL. Therapeutic anti-CD3 monoclonal antibodies: from bench to bedside. Immunotherapy. 2016 Jul;8(8):889-906. doi: 10.2217/imt-2016-0049. Epub 2016 May 10. PMID 27161438
- [Background] Krasemann S, Madore C, Cialic R, Baufeld C, Calcagno N, El Fatimy R, Beckers L, O'Loughlin E, Xu Y, Fanek Z, Greco DJ, Smith ST, Tweet G, Humulock Z, Zrzavy T, Conde-Sanroman P, Gacias M, Weng Z, Chen H, Tjon E, Mazaheri F, Hartmann K, Madi A, Ulrich JD, Glatzel M, Worthmann A, Heeren J, Budnik B, Lemere C, Ikezu T, Heppner FL, Litvak V, Holtzman DM, Lassmann H, Weiner HL, Ochando J, Haass C, Butovsky O. The TREM2-APOE Pathway Drives the Transcriptional Phenotype of Dysfunctional Microglia in Neurodegenerative Diseases. Immunity. 2017 Sep 19;47(3):566-581.e9. doi: 10.1016/j.immuni.2017.08.008. PMID 28930663
- [Background] Keymeulen B, Vandemeulebroucke E, Ziegler AG, Mathieu C, Kaufman L, Hale G, Gorus F, Goldman M, Walter M, Candon S, Schandene L, Crenier L, De Block C, Seigneurin JM, De Pauw P, Pierard D, Weets I, Rebello P, Bird P, Berrie E, Frewin M, Waldmann H, Bach JF, Pipeleers D, Chatenoud L. Insulin needs after CD3-antibody therapy in new-onset type 1 diabetes. N Engl J Med. 2005 Jun 23;352(25):2598-608. doi: 10.1056/NEJMoa043980. PMID 15972866
- [Background] Ilan Y, Zigmond E, Lalazar G, Dembinsky A, Ben Ya'acov A, Hemed N, Kasis I, Axelrod E, Zolotarov L, Klein A, El Haj M, Gandhi R, Baecher-Allan C, Wu H, Murugaiyan G, Kivisakk P, Farez MF, Quintana FJ, Khoury SJ, Weiner HL. Oral administration of OKT3 monoclonal antibody to human subjects induces a dose-dependent immunologic effect in T cells and dendritic cells. J Clin Immunol. 2010 Jan;30(1):167-77. doi: 10.1007/s10875-009-9323-7. Epub 2009 Sep 16. PMID 19756989
- [Background] Faridar A, Thome AD, Zhao W, Thonhoff JR, Beers DR, Pascual B, Masdeu JC, Appel SH. Restoring regulatory T-cell dysfunction in Alzheimer's disease through ex vivo expansion. Brain Commun. 2020 Jul 20;2(2):fcaa112. doi: 10.1093/braincomms/fcaa112. eCollection 2020. PMID 32954348
- [Background] Dansokho C, Ait Ahmed D, Aid S, Toly-Ndour C, Chaigneau T, Calle V, Cagnard N, Holzenberger M, Piaggio E, Aucouturier P, Dorothee G. Regulatory T cells delay disease progression in Alzheimer-like pathology. Brain. 2016 Apr;139(Pt 4):1237-51. doi: 10.1093/brain/awv408. Epub 2016 Feb 1. PMID 26912648
- [Background] Colonna M, Butovsky O. Microglia Function in the Central Nervous System During Health and Neurodegeneration. Annu Rev Immunol. 2017 Apr 26;35:441-468. doi: 10.1146/annurev-immunol-051116-052358. Epub 2017 Feb 9. PMID 28226226
- [Background] Ciccocioppo F, Lanuti P, Pierdomenico L, Simeone P, Bologna G, Ercolino E, Buttari F, Fantozzi R, Thomas A, Onofrj M, Centonze D, Miscia S, Marchisio M. The Characterization of Regulatory T-Cell Profiles in Alzheimer's Disease and Multiple Sclerosis. Sci Rep. 2019 Jun 19;9(1):8788. doi: 10.1038/s41598-019-45433-3. PMID 31217537
- [Background] Butovsky O, Jedrychowski MP, Moore CS, Cialic R, Lanser AJ, Gabriely G, Koeglsperger T, Dake B, Wu PM, Doykan CE, Fanek Z, Liu L, Chen Z, Rothstein JD, Ransohoff RM, Gygi SP, Antel JP, Weiner HL. Identification of a unique TGF-beta-dependent molecular and functional signature in microglia. Nat Neurosci. 2014 Jan;17(1):131-43. doi: 10.1038/nn.3599. Epub 2013 Dec 8. PMID 24316888
- [Background] Baek H, Ye M, Kang GH, Lee C, Lee G, Choi DB, Jung J, Kim H, Lee S, Kim JS, Lee HJ, Shim I, Lee JH, Bae H. Neuroprotective effects of CD4+CD25+Foxp3+ regulatory T cells in a 3xTg-AD Alzheimer's disease model. Oncotarget. 2016 Oct 25;7(43):69347-69357. doi: 10.18632/oncotarget.12469. PMID 27713140
- [Background] Alves S, Churlaud G, Audrain M, Michaelsen-Preusse K, Fol R, Souchet B, Braudeau J, Korte M, Klatzmann D, Cartier N. Interleukin-2 improves amyloid pathology, synaptic failure and memory in Alzheimer's disease mice. Brain. 2017 Mar 1;140(3):826-842. doi: 10.1093/brain/aww330. PMID 28003243
- See also: AmyvidTM Package Insert, 2012. United States Package Insert for florbetapir F18 Injection . — https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/202008s000lbl.pdf